CLINICAL TRIAL: NCT04946786
Title: Role of Clinical, Biochemical and Body Composition Analysis in Assessment of Steatosis in Patients With Non Alcoholic Fatty Liver Disease
Brief Title: Clinical, Biochemical and Body Composition Analysis in Assessment of Steatosis in Non Alcoholic Fatty Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Wafaa Gamal Mohamed, priciple investigator, Sohag University
Other Study IDs: Soh-Med-21-06-13
Record Dates: First submitted 2021-06-13; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Non-alcoholic Fatty Liver Disease NAFLD
Keywords: Non-alcoholic fatty liver disease NAFLD

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Laboratory investigations, pelvi-abdominal US, fibroscan, and in body analysis — 1. Complete history taking.
  2. Thorough clinical examination :Assessing for buffalo hump, double chin, acanthosis nigricans, skin tags or acrochordon and xanthelasma and anthropometric measurements as measuring height "m", weight "Kg", waist circumference (WC) "Cm", hip circumference (HC) "Cm".
  3. Pelvi-abdominal ultrasound. 4. Fibroscan examination will be done for all subjects to assess steatosis by measuring the CAP score.
  5. Body composition analysis: to detect water, muscle and fat percentage in the body.
  6. Laboratory investigations:All samples wil be analyzed for fasting blood glucose (FBG), and post-prandial (2hrs after meals) blood glucose, total cholesterol (TC), triglycerides (TG), high-density lipoprotein cholesterol (HDL-C), very low-density lipoprotein (VLDL-C), alkaline phosphatase (ALK), aspartate transaminase (AST),alanine transaminase (ALT).
  • Fasting insulin levels will be measured using ELISA kits

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) includes a spectrum of liver disorders characterized by accumulation of hepatic fat in absence of significant alcohol consumption (<20 gm/day) and other causes of liver diseases. It is the most common cause of asymptomatic elevation of liver enzymes worldwide (Marchesini et al., 2003).

Unfortunately, to date, existing non- or minimally invasive biomarkers are inadequate. While a number of non- or minimally invasive tests are able to rule out ﬁbrosis or cirrhosis, no single test to identify steatosis, to early diagnose NASH, or to predict the disease progression is available. Moreover, specialized, combined tests are required to assess treatment response in clinical trials on emerging compounds (Piazzolla and Mangia, 2020).

Among minimally invasive tools, plasma biomarkers and composite scores defined as "wet biomarkers" are commonly used. For example, fasting insulin level and its use in measurement of insulin resistance, Lipid Accumulation Product (LAP) score (Bedogni et al., 2010), the NAFLD Liver Fat Score (NLFS) (Kontronen et al., 2009), Hepatic Steatosis Index (HSI) (Lee et al., 2010), controlled attenuation parameter (CAP) measurement by fibroscan (Piazzolla and Mangia, 2020). Recent studies have shown that CAP signiﬁcantly correlates with the percentage of steatosis and steatosis grade and that median CAP is higher among patients with signiﬁcant steatosis (Sasso et al., 2012 & Karlas et al., 2017).

The prevalence of NAFLD is 80-90% in obese, 30-50% in patients with diabetes and up to 90% in patients with hyperlipidemia (Abenavoli et al., 2014)

Central obesity or visceral fat (VF) (determined by waist circumference (WC)) is defined as the presence of excess fat in the abdomen, and this type of obesity is often associated with the development and progression of NAFLD or more advanced forms of liver disease (Abenavoli et al., 2016). Thus, measurement of body composition rather than BMI may be helpful in the prediction of NAFLD (Milić et al., 2014 and Abenavoli et al., 2016)

There is a growing need to assess the steatosis in NAFLD patients using minimally invasive tools.

ELIGIBILITY:
Inclusion criteria:

* Adult subjects with bright liver by abdominal ultrasound will be recruited.
* The diagnosis will be based on CAP score result measured by Fibroscan.

Exclusion criteria:

* Alcohol consumption.
* Patients with other liver diseases as acute and chronic viral hepatitis, autoimmune hepatitis, primary biliary cirrhosis, drug-induced hepatitis.
* Decompensated liver disease.
* Other end organ failure.
* Pregnancy.
* Patients on statins or fenofibrate.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients: A total of 80 adult subjects will be included.
  Inclusion criteria:
  Adult subjects with bright liver by abdominal ultrasound will be recruited for the study. The diagnosis will be based on CAP score result measured by Fibroscan.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
studying anthropometric measurements of NAFLD cases. | 2 years
  -study anthropometric measurements.
measurement of steatosis by fibroscan examination | 2 years
  Fibroscan examination measuring control attenuation parameter "CAP score"
body muscle percentage | 2 years
  measurement of body muscle percentage
body fat percentage. | 2 years
  measurement of body fat percentage
measurement of body water percentage. | 2 years
  measurement of body water percentage.
measuring serum cholesterol | 2 years.
  measuring serum cholesterol by mg/ dl.
measuring serum triglycerides. | 2 years.
  measuring serum triglycerides by mg/ dl.
measuring serum insulin level. | 2 years.
  measuring of serum insulin level using ELISA kits

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Abenavoli L, Di Renzo L, De Lorenzo A. Body Composition and Non-alcoholic Fatty Liver Disease. J Lifestyle Med. 2016 Mar;6(1):47-8. doi: 10.15280/jlm.2016.6.1.47. Epub 2016 Mar 31. No abstract available. PMID 27358840
- [Background] Abenavoli L, Milic N, Peta V, Alfieri F, De Lorenzo A, Bellentani S. Alimentary regimen in non-alcoholic fatty liver disease: Mediterranean diet. World J Gastroenterol. 2014 Dec 7;20(45):16831-40. doi: 10.3748/wjg.v20.i45.16831. PMID 25492997
- [Background] Amato MC, Giordano C, Galia M, Criscimanna A, Vitabile S, Midiri M, Galluzzo A; AlkaMeSy Study Group. Visceral Adiposity Index: a reliable indicator of visceral fat function associated with cardiometabolic risk. Diabetes Care. 2010 Apr;33(4):920-2. doi: 10.2337/dc09-1825. Epub 2010 Jan 12. PMID 20067971